CLINICAL TRIAL: NCT01234194
Title: Changes in the Composite Variability Index in Response to Different Remifentanil Concentrations and Standardized Painful Stimuli.
Brief Title: Composite Variability Index and Propofol Remifentanil Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Richard Klaus Ellerkmann / M.D., University of Bonn
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CVI_2010
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-09

CONDITIONS: Measure of Nociception
Keywords: Composite Variability Index; Bispectral Index; Electromyography; Nociception; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: rising remifentanil concentrations
- Group 2 (Active Comparator)
  Interventions: Drug: falling remifentanil concentrations

INTERVENTIONS:
Drug: rising remifentanil concentrations — remifentanil effect-compartment concentrations 0,1,2,3 ng/ml
  Arms: Group 1
Drug: falling remifentanil concentrations — remifentanil effect-compartment concentrations 3, 2, 1, 0 ng/ml
  Arms: Group 2

SUMMARY:
The purpose of the study is to determine if the new Composite Variability Index (CVI) is capable of detecting changing effect compartment concentrations of remifentanil. In addition, it is planed to detect if the change in CVI in response to a standardized painful stimulus is dose-dependent.

DETAILED DESCRIPTION:
On the day of surgery, patients receive anesthesia by propofol infusion. As soon as the patient is unresponsive und unconscious (BIS 40-60) and a steady state is achieved, a standardized painful stimulus is applied by electrical stimulation of the ulnar nerve (tetanic stimulation [70 mA], 30 seconds, 50 Hz) in group 1. Thereafter remifentanil is infused to an effect compartment concentration target of 1 ng/ml. The standardized stimulus is applied again as the remifentanil target is reached. This procedure is repeated with remifentanil targets of 2 ng/ml and 3ng/ml. In group 2 remifentanil is targeted to effect compartment concentrations of 3 ng/ml followed by 2,1, and 0 ng/ml.

After measuring the effect of the last painful stimulus the patient is intubated for surgery. Throughout the study the Composite Variability Index and standard monitoring is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical procedure in general anesthesia

Exclusion Criteria:

* Pregnancy, drug abuse, cardiac arrhythmia, obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Prediction Probability of CVI versus remifentanil effect compartment concentration and versus movement after painful stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Ellerkmann, M.D., Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany